CLINICAL TRIAL: NCT00514423
Title: How Can Rehospitalisations of Patients With Schizophrenia be Avoided? A Comparison Between Different Compliance Programs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01GL0509; ISRCTN19638644
Record Dates: First submitted 2007-08-09; First posted 2007-08-10 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Schizophrenia; Schizoaffective Disorder
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Control Groups

ARMS (4):
- 2 (Experimental): Psychoeducation by peer-moderators
  Interventions: Other: Psychoeducation by peer-moderators
- 1 (Experimental): Psychoeducation by professionals
  Interventions: Other: Psychoeducation by professonals
- 3 (Experimental): Video-education
  Interventions: Other: Video-education
- 4 (Placebo Comparator): Control group
  Interventions: Other: Noneducational video group (control group)

INTERVENTIONS:
Other: Psychoeducation by professonals
  Arms: 1
Other: Psychoeducation by peer-moderators
  Arms: 2
Other: Video-education
  Arms: 3
Other: Noneducational video group (control group)
  Arms: 4

SUMMARY:
Participation in one of the three interventions psychoeducation by professionals, psychoeducation by peer-moderators, or video-education can reduce the rehospitalisation rate of patients with schizophrenia compared to a control group.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia or schizoaffective disorder (ICD-10)
* Age 18 to 67 years
* Hospitalised or treated in day care clinic

Exclusion Criteria:

* More than 12 months of hospitalisation within the last two years
* Substance-dependency (principal diagnosis)
* Mental retardation ICD-10 Chapter F70-79
* Fluency of German language not given

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Estimated)
Dates: Start 2006-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rehospitalisation rate

SECONDARY OUTCOMES:
Rehospitalisation days
Resulting costs per patient
Compliance
Knowledge of illness
Attitude towards illness
Quality of life
Satisfaction with treatment
Duration of consultation time
Dealing with mental illness

CONTACTS AND LOCATIONS:
Overall Officials: Werner Kissling, MD, Principal Investigator — Technical University of Munich
Locations (1):
- Klinik und Poliklinik für Psychiatrie und Psychotherapie am Klinikum rechts der Isar der Technischen Universität München, München, Germany